CLINICAL TRIAL: NCT05998629
Title: Skin-interfaced Colorimetric Bifluidic Sweat Sensor Device for the Diagnosis of Cystic Fibrosis (CF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Robert Vender, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 7772
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
Keywords: Sweat Chloride Test; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Comparison of sweat chloride measure using standard of care versus experimental device in both control and cystic fibrosis subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy control subjects experimental device (Experimental): a skin-interfaced colorimetric bifluidic sweat device with two synchronous channels for healthy control subjects
  Interventions: Device: a skin-interfaced colorimetric bifluidic sweat device with two synchronous channels
- Healthy control subjects standard of care (Active Comparator): standard clinical laboratory procedures routinely performed in the Clinical Laboratory at Penn State Health Milton S. Hershey Medical Center (PSH-HMC), Hershey, PA for measurement of sweat chloride concentrations for healthy control subjects
  Interventions: Other: Standard of Care laboratory procedure for measurement of sweat
- Cystic Fibrosis Subjects experimental device (Experimental): a skin-interfaced colorimetric bifluidic sweat device with two synchronous channels for cystic fibrosis subjects
  Interventions: Device: a skin-interfaced colorimetric bifluidic sweat device with two synchronous channels
- Cystic Fibrosis Subjects standard of care (Active Comparator): standard clinical laboratory procedures routinely performed in the Clinical Laboratory at Penn State Health Milton S. Hershey Medical Center (PSH-HMC), Hershey, PA for measurement of sweat chloride concentrations for cystic fibrosis subjects
  Interventions: Other: Standard of Care laboratory procedure for measurement of sweat

INTERVENTIONS:
Device: a skin-interfaced colorimetric bifluidic sweat device with two synchronous channels — a skin-interfaced colorimetric bifluidic sweat device with two synchronous channels
  Arms: Cystic Fibrosis Subjects experimental device; Healthy control subjects experimental device
Other: Standard of Care laboratory procedure for measurement of sweat — a skin-interface sweat measurement using a smart-watch type device
  Arms: Cystic Fibrosis Subjects standard of care; Healthy control subjects standard of care

SUMMARY:
Cystic fibrosis (CF) is a multisystem autosomal recessive inherited disease affecting approximately 75,000 individuals in USA. The sweat chloride (Cl) test remains the gold standard for diagnosis of CF but still has a number of limitations. The objectives of this study are: 1)To evaluate a skin-interfaced colorimetric bifluidic sweat device with two synchronous channels as a potential low-cost but potentially accurate test to diagnoses cystic fibrosis (CF) and 2) To evaluate measurements of sweat chloride (Cl) using this same system in comparison to the standard clinical laboratory procedures routinely performed in the Clinical Laboratory at Penn State Health Milton S. Hershey Medical Center (PSH-HMC), Hershey, PA for assessment of the diagnosis of CF. This is a single institution study performed solely at PSH-HMC. Study participants will include 1) adults 18 years of age or older capable of providing signed and dated informed consent, 2) subjects with an established known diagnosis of cystic fibrosis (CF) or healthy volunteers, and 3) able to understand and speak English language. Exclusion criteria include: 1) any medical condition or disorder known to potentially interfere with accurate measurements of sweat chloride and 2) inability to understand and speak the English language. Cystic Fibrosis (CF) subjects will be identified from the population of eligible patients receiving medical care at Penn State Health- Milton S. Hershey Medical Center (PSH-HMC). Healthy donor volunteers will be recruited from various members of the PSH-HMC CF clinical care team, members of the Division of Allergy, Pulmonary and Critical Care (both faculty and trainees) at PSH-HMC, and PSU-University Park research team. The total projected number of combined enrolled subjects is 30. This is a single day single time study that will require approximately 60 minutes of subject participation. Potential risks include a) side effects from pilocarpine iontophoresis sweat test collection (pain, skin discomfort, blisters, rarely burns and b) loss of confidentiality. There will be no cost to subjects for study participation. There will be no reimbursement financially for study participation. There is no benefit to subjects for study participation. There is the potential benefit to medical science via identification of improved method to accurately measure sweat chloride for diagnosis of CF.

DETAILED DESCRIPTION:
Background: Cystic fibrosis (CF) is a multisystem autosomal recessive inherited disease affecting approximately 75,000 individuals in USA. The sweat chloride (Cl) test remains the gold standard for diagnosis of CF but still has a number of limitations including 1) common inability to recover enough sweat volume for test accuracy, termed "quantity not sufficient" limitation, 2) difficulty of performing in young children and infants, 3) absence of point of care (POC) simplicity and need to schedule prolonged (> 1 hour) appointment with high resource and personnel utilization, and 4) still a range of values without one specific diagnostic cut-off measurement thus creating sweat Cl classifications of negative (normal), indeterminant, and positive (diagnostic). Multiple publications already exist validating the use of POC skin-interfaced micro fluidic colorimetric systems in attempts to overcome these limitations of the still standard of care macroduct sweat collection and analysis system. The current proposed investigational diagnostic (not therapeutic) device introduces a skin-interfaced colorimetric bifluidic sweat collection and analyses device with two synchronous channels to quantify sweat rate and biomarkers (for this study Cl) in real-time, even during uncertain sweat conditions and activities. This proposed bifluidic system could provide accurate analysis of biomarkers (including Cl) based upon instantaneous sweat rate. For consistent of data accrual and analyses in this proposed study, for both methods of sweat collection pilocarpine iontophoresis will be the method of sweat stimulation. This skin-interfaced colorimetric bifluidic sweat device with two synchronous channels device is a closed system design to reduce evaporation and resists contamination from the external environment. This low-cost yet highly accurate device provides opportunities for clinical sweat analysis and disease screening in remote and low-resource settings which is currently non-existent with standard clinical measurements of sweat Cl. In addition, this device can be easily adapted for other biomarkers, when corresponding colorimetric reagents are exploited.

Inclusion Criteria: 1) Adults 18 years of age or older capable of providing signed and dated informed consent, 2) Subjects with an established know diagnosis of cystic fibrosis (CF) or healthy volunteers, 3) Competent to understand written and spoken English language.

Exclusion Criteria: Participants receiving medications or with known disorders that can cause errors in sweat test analysis. Common causes of potential error inducing factors in sweat test determination include Lithium therapy, mineralocorticoid hormone therapy, adrenal insufficiency, glycogen storage diseases, hypothyroidism, hypoparathyroidism, nephrogenic diabetes insipidus, G6PD deficiency, ectodermal dysplasia, or any skin or soft tissue disorders that could affect obtaining the necessary volume and quality of sweat. Non-English-speaking subjects will be excluded.

Study Design: This is a single institution study to be performed entirely at the Penn State Health Milton S. Hershey Medical Center (PSH-HMC), Hershey, PA. This is only a single day, single time study, i.e. VISIT 1 and DAY 1 ONLY. The study involves minimal risk. There is no anticipated benefit to subjects for study participation. Total subject participation time will be approximately 60 minutes, after which subjects' participation will end. The total combined estimated enrollment for both health volunteer subjects and CF subjects will be 30. Two sweat chloride samples and measurements as per study procedures will be obtained simultaneously from both arms using pilocarpine iontophoresis.

Study Procedures: 1) PSH-HMC Clinical Laboratory Department of Pathology SOP dated 14-Nov-2022 "Macroduct Sweat Collection" will be complied for attainment of the sample for which sweat chloride will be measured at PSH-HMC. The site for this procedure is Suite 520 at the University Physicians Center, Hershey, PA. After completion of pilocarpine iontophoresis and following collection of sweat specimens inside the macroduct tubing, the sweat will then be eluted and analyzed separately. PSH-HMC sample chloride biochemical analyses: a) add reached 12 μL as indicated in the microfluidic device. The measured color change distance will be used to determine the chloride concentration according to the linear relationship.2N nitric acid and s-Diphenylcarbazone, b) rinse with 0.005N mercuric nitrate and titrate to very light purple color and record volume of mercuric nitrate, c) prepare control standards, d) calculate the chloride result using the EXCEL calculation template.

2) PSU-UP sample chloride biochemical analyses: The real-time quantification of sweat rate and chloride will also be pursued with a skin-interfaced colorimetric microfluidic sweat device developed at Penn State University- University Park, PA (PSU-UP). In brief, the skin of the human subjects will first be washed with soap and water and dried with disposable paper. The device will be attached to the skin near pilocarpine iontophoresis. The experiment will end after the collected sweat.

Risks: 1) The attainment of the sweat chloride sample for analyses involves only minimal risk. Obtaining a sweat chloride sample entails approximately 45-60 minutes for volume collections plus as per the standard process of pilocarpine iontophoresis (which is the chemical and electrical process used to stimulate the production of sufficient volumes of sweat) for approximately 5-10 minutes. CF patients may have had this sweat chloride test performed at an early age as part of their diagnostic evaluation for CF. During this time period of collection a electrical charge will be delivered via a battery device to the two electrodes attached to the skin of both forearms which may cause discomfort such as numbness, tingling, pins and needles sensation or actual pain, and is expected to resolve with termination of tests without any expectation of long term sequelae or injury. If such discomfort becomes excessive or intolerant as per study participant, the process will be terminated. When the pilocarpine iontophoresis procedure is completed the skin under the gel pads usually looks red and puffy. Occasionally small whitish blisters can appear. Both conditions fade quickly and usually disappear without two hours. Very rarely small burns or blisters can occur. This happens in less than 1 in 50,000 patients. Two samples will be obtained from separate arms simultaneously at a single timepoint. 2) The recovery of any private health related information always creates the potential of risk of disclosing this information beyond the intent of this research study. In accordance with PSH-HMC and Federal guidelines and policies , all precautions will be taken to avoid this risk including the "coding" of personal identifiable information and protected health information (including name, medical record number [if available], age, date of birth, gender, race, medications) and the security of any information linking this code to personal health and personal identifiable information being secured in a locked office of Dr. Vender in Biomedical Research Building (C5860F).

ELIGIBILITY:
Inclusion Criteria:

* adults 18 years of age or older capable of providing signed and dated informed consent,
* subjects with an established known diagnosis of cystic fibrosis (CF) or healthy volunteers,
* able to understand and speak English language.

Exclusion Criteria:

* any medical condition or disorder known to potentially interfere with accurate measurements of sweat chloride
* inability to understand and speak the English language.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Sweat chloride concentration using standard of care lab assessment | Single point in time measurement 60 minutes after device attachment
  Sweat chloride concentration in mmol/L

SECONDARY OUTCOMES:
Sweat chloride concertation using skin-interfaced colorimetric device | Single point in time measurement 60 minutes after device attachment
  Sweat chloride concentration in mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No